CLINICAL TRIAL: NCT01517698
Title: A Randomized, Double-blind, 12-week, Parallel Group, Placebo-controlled Study of Efficacy and Safety of RO4917523 in Patients With Fragile X Syndrome.
Brief Title: A Study of RO4917523 in Patients With Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP27936
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — 2-chloro-4-(1-(4-fluorophenyl)-2,5-dimethyl-1H-imidazol-4-ylethynyl)pyridine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- RO4917523 0.5 mg (Experimental)
  Interventions: Drug: RO4917523 0.5 mg
- RO4917523 1.5 mg (Experimental)
  Interventions: Drug: RO4917523 1.5 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — placebo to RO4917523 orally once a day for 12 weeks
  Arms: Placebo
Drug: RO4917523 0.5 mg — 0.5 mg orally once a day for 12 weeks
  Arms: RO4917523 0.5 mg
Drug: RO4917523 1.5 mg — 1.5 mg orally once a day for 12 weeks
  Arms: RO4917523 1.5 mg

SUMMARY:
This multi-center, randomized, double-blind, placebo-controlled, parallel-group study will investigate the efficacy and safety of RO4917523 in adolescent and adult patients with fragile X syndrome. Patients will be randomized to receive oral doses of 0.5 mg or 1.5 mg of RO4917523, or matching placebo once daily. The anticipated time on study treatment is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult and adolescent patients, 14-50 years of age
* Diagnosis of fragile X syndrome with a confirmed fragile X mental retardation 1 (FMR1) full mutation and qualifying scores on the Aberrant Behavior Checklist (ABC) and CGI-S
* Patients must agree to either remain completely abstinent or to use two effective contraceptive methods during and 3 weeks after the study

Exclusion Criteria:

* Previous treatment with another metabotropic glutamate (mGLU) receptor antagonist within 18 months or with RO4917523
* Participation in a clinical trial involving an investigational (unapproved) drug within 3 months or 5 times the half-life (whichever is longer) before start of this study
* Any uncontrolled, unstable clinically significant psychiatric condition other than fragile X syndrome
* History of suicidal behavior

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 185 (Actual)
Dates: Start 2012-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety Depression and Mood Scale (ADAMS) total score | 12 weeks
Safety (incidence of adverse events) | 12 weeks

SECONDARY OUTCOMES:
Change in Social Responsiveness Scale (SRS) | 12 weeks
Change in Clinical Global Impressions Scale - Improvement (CGI-I) | 12 weeks
Change in Clinical Global Impressions Scale - Severity of Illness (CGI-S) | 12 weeks
Change in Aberrant Behavior Checklist total score | 12 weeks
Change in Aberrant Behavior Checklist factor scores | 12 weeks
Change in Anxiety Depression and Mood Scale (ADAMS) factor scores | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (48):
- United States (20):
  - Phoenix, Arizona
  - Long Beach, California
  - Sacramento, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Decatur, Georgia
  - Chicago, Illinois
  - Iowa City, Iowa
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Worcester, Massachusetts
  - New York, New York
  - Staten Island, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Media, Pennsylvania
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Seattle, Washington
- Argentina (2):
  - Bahía Blanca
  - Caba
- Canada (2):
  - Brampton, Ontario
  - Sherbrooke, Quebec
- Chile (2):
  - Santiago
  - Valparaíso
- France (7):
  - Bordeaux
  - Bron
  - Dijon
  - Marseille
  - Montpellier
  - Paris
  - Tours
- Mexico (2):
  - Aguascalientes
  - México
- Lima, Peru
- Spain (5):
  - San Cugat Del Valles, Barcelona
  - Donostia / San Sebastian, Guipuzcoa
  - Madrid, Madrid
  - Torremolinos, Malaga
  - El Palmar. Murcia, Murcia
- Gothenburg, Sweden
- United Kingdom (6):
  - Belfast
  - Dundee
  - Edinburgh
  - Glasgow
  - London
  - Manchester